CLINICAL TRIAL: NCT00453778
Title: A Study to Investigate the Effect of Inhaled Fluticasone Propionate on the Bronchial Responsiveness to Leukotriene D4 in Asthmatics Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FMS40273
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Asthma; Mild Asthma
Keywords: mild asthma; FLIXOTIDE; methacholine; bronchial challenge; leukotriene D4
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: FLIXOTIDE Diskus 500 mcg (Fluticasone Propionate)

SUMMARY:
Investigate if asthmatics treated with FLIXOTIDE (FP) 500 mcg BID during 14 days get reduced bronchial reactivity after inhalation of Leukotriene D4. Two 14 days treatment periods where patients received FP 500 MCG BID and placebo. Washout at least 21 days between treatments. Bronchial challenge with methacholine and Leukotriene D4 were performed before the start of each treatment period and on treatment days 13 and 14 respectively.

ELIGIBILITY:
Inclusion:

* Diagnosed history of asthma
* Non smoker last two years
* < 5 pack years
* FEV1 >70% of predicted
* Mild and stable asthma
* Only using short acting b2-agonist as rescue for the last 4 weeks
* Have a history of atopy.

Exclusion:

* Any significant respiratory disease, other than asthma
* Subjects with seasonal asthma may not be included if they are in their season
* Use of oral or inhaled glucocorticosteroid for the last 3 months and long-acting or oral b2-agonists, anticholinergic bronchodilators, cromones, antihistamines, theophyllines and antileukotrienes within two weeks
* Upper or lower RTI within 6 weeks
* Evidence of any disease that in the investigators mind would affect the results of the study
* Participating in another study within 4 weeks
* Females who are pregnant, intend to be or who are lactating
* Methacholine PD20 > 454mcg
* Negative scin prick test

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14
Dates: Start 2002-11; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
LTD4 PC20

SECONDARY OUTCOMES:
Shift in methacholine PD20

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline